CLINICAL TRIAL: NCT03401489
Title: Program to Avoid Cerebrovascular Events Through Systematic Electronic Tracking and Tailoring of an Eminent Risk-factor
Brief Title: PACESETTER: Program to Avoid Cerebrovascular Events Through Systematic Electronic Tracking and Tailoring of an Eminent Risk-factor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study delays and ran out of funding
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: University of South Carolina (Other); Medical University of South Carolina (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Bruce Ovbiagele, Chief of Staff, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00070627; 5R01MD012441-05 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure; Hypertension; Mhealth
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PACESETTER (Experimental): Participants in the PACESETTER arm received a multicomponent, mHealth-enabled self-management program designed to improve post-stroke blood-pressure control. Each participant was provided a Bluetooth-enabled UA-767Plus BT home blood-pressure monitor, a Vaica electronic medication tray that emitted visual and auditory reminders, and the PACESETTER smartphone app.
  The app delivered instructional videos, enabled automatic transmission of BP and adherence data to a secure server, and generated tailored SMS messages based on self-determination-theory constructs of competence and autonomous regulation. Participants also received twice-weekly educational text messages regarding hypertension and stroke prevention, medication adherence, and communication with clinicians.
  Bi-weekly adherence and BP summaries were sent to study physicians to guide medication adjustments. Study coordinators contacted participants monthly to ensure device functioning and collect follow-up data.
  Interventions: Device: PACESETTER
- Healthy Lifestyle Intervention Group (No Intervention): General lifestyle SMS matched in frequency and length to the intervention; monthly follow-ups; no devices, adherence monitoring, or physician-directed feedback.

INTERVENTIONS:
Device: PACESETTER — Patients will be given a Vaica electronic pill tray & blue-toothed UA-767 Plus BT BP device and the PACESETTER app installed on their smart phone for automatic relay of BP data. The Vaica tray emits a blinking light for 30 minutes when it is time to take the meds. If the compartment is not opened and emptied, an intermittent chime ensues for 30 minutes. If the compartment is not opened and emptied, the subject /caregiver receives an automated SMS. PACESETTERs will be given a questionnaire. Responses will be used to generate personalized motivational & reinforcement messages guided by self-determination theory constructs of competence & autonomous regulation. In addition to personalized messages, PACESETTERs will receive text messages 2 times per week on HTN/stroke facts, importance of med adherence, and tips on expressing questions/concerns with a physician. We will calculate medication possession ratios, on all subjects' HTN medications at each evaluation.
  Arms: PACESETTER

SUMMARY:
Program to Avoid Cerebrovascular Events through Systematic Electronic Tracking and Tailoring of an Eminent Risk-factor (PACESETTER) aims to assess the incorporation of its stroke intervention into 2 safety net/academic health systems in a given US state especially burdened by stroke, thereby enhancing knowledge about the complexity of stroke interventions, and especially the nature of the challenges encountered in low resource settings and for populations traditionally underrepresented in research. Altogether, the intervention, if proven implementable and effective, may eventually be exported to other medically underserved populations in the US beyond SC as a feasible model of post-stroke management.

ELIGIBILITY:
Inclusion Criteria:

* African American or non-Hispanic white
* history of stroke (within six months of symptom onset)
* uncontrolled HTN (SBP ≥ 130 mmHg at the last clinical encounter post-stroke prior to recruitment)
* owning a smartphone with a data plan
* able to take their own BP and self-administer medications.

Exclusion Criteria:

* Any condition that would limit participation in follow up assessments including severe cognitive impairment/dementia

  * severe global disability (modified Rankin Score ≥ 3)
  * BMI> 40kg/m^2
  * Not being able to speak, hear, or understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NCIRE, San Francisco, California
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - Regional Medical Center: Orangeburg Hospital, Orangeburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wabnitz AM, Chandler J, Treiber F, Sen S, Jenkins C, Newman JC, Mueller M, Tinker A, Flynn A, Tagge R, Ovbiagele B. Program to Avoid Cerebrovascular Events through Systematic Electronic Tracking and Tailoring of an Eminent Risk factor: Protocol of a RCT. J Stroke Cerebrovasc Dis. 2021 Aug;30(8):105815. doi: 10.1016/j.jstrokecerebrovasdis.2021.105815. Epub 2021 May 27. PMID 34052785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stroke survivors with uncontrolled systolic hypertension were recruited from two safety-net health systems in South Carolina (MUSC and USC) between July 2020-February 2024. Potential participants were identified through EMR review and clinic screening. Recruitment ended at 60% of target due to COVID-19 disruptions and loss of funding. A total of 120 patients were enrolled and randomized 1:1.
Pre-assignment Details: We assessed 200 individuals for eligibility; 80 did not meet inclusion criteria and declined participation, leaving 120 ischemic stroke patients with uncontrolled systolic hypertension who were randomized (60 intervention, 60 usual care). Randomization was stratified by race and site using permuted blocks within REDCap. All participants provided written informed consent prior to assignment
Groups:
- PACESETTER: Participants received a multicomponent mHealth-enabled self-management program. The intervention included a Bluetooth-enabled UA-767Plus BT home blood pressure monitor, an electronic medication pill tray (Vaica), and the PACESETTER smartphone app. The app provided instructional videos, automated relay of BP and adherence data to a secure server, and tailored SMS reminders and motivational messages. Biweekly adherence and BP summary reports were sent to study physicians to guide medication adjustments.
- Healthy Lifestyle Intervention Group: Participants continued standard post-stroke hypertension care. To balance contact frequency, they received general lifestyle SMS messages (not related to BP or medication adherence) matched in frequency and length to the intervention arm. Monthly phone calls from study staff confirmed follow-up and health encounters. No electronic devices, adherence monitoring, or physician-directed feedback were provided.
Period: Overall Study
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group
Started | 60 | 60
Completed | 26 | 21
Not Completed | 34 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, Continuous: Mean ± SD
  years | 61.1 (10.2) | 59.7 (10.9) | 60.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Male/Female
  Participants
    Female | 25 | 27 | 52
    Male | 35 | 33 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 38 | 77
  White | 21 | 22 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants] — South Carolina, USA
  Participants
    United States | 60 | 60 | 120
Modified Rankin Score (mRS) [Mean (Standard Deviation); unit: units on a scale] — The Modified Rankin Scale (mRS) measures the degree of disability or dependence in daily activities after a stroke. The total score ranges from 0 to 6, where 0 = no symptoms (best outcome) and 6 = death (worst outcome). Lower scores indicate better functional outcomes. Scores were assessed by a blinded outcomes assessor at baseline.
  units on a scale | 1.8 (.09) | 1.9 (.08) | 1.85 (0.85)
Baseline DBP (mmHg) [Mean (Standard Deviation); unit: mmHg] — Baseline Diastolic Blood Pressure
  mmHg | 85.7 (12.8) | 88 (10.1) | 86.9 (11.5)
Number of Daily Medications ≥ 5 [Count of Participants; unit: Participants] | 43 | 39 | 82
Insurance Status [Count of Participants; unit: Participants]
  Private | 24 | 24 | 48
  Medicare/Medicaid | 23 | 17 | 40
  Both | 9 | 11 | 20
  No insurance | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Systolic Blood Pressure <130 mmHg at 12 Months
Description: Clinic systolic blood pressure (SBP) was measured at 12 months after randomization. The proportion of participants in each arm achieving SBP <130 mmHg was calculated.
Time Frame: 12 months
Population: Participants dropped out and in addition, the study was ended prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group
Number analyzed (Participants) | 32 | 40
Participants | 15 | 17
Statistical Analysis 1: Comparison: PACESETTER vs Healthy Lifestyle Intervention Group; Comparison between PACESETTER and control arms at 12 months for proportion of participants with SBP <130 mmHg using a generalized linear mixed model (GLMM) with logit link. Model included baseline SBP, site, and race as covariates; Test type: Superiority; p = 0.822, Mixed Models Analysis — Significance threshold was α=0.05, two-sided. No adjustment for multiple comparisons; Generalized linear mixed models were also run for sensitivity analyses, adjusting for baseline SBP, site, and race; Odds Ratio (OR) = 0.99, 95% CI 2-sided [.36 to 2.72] — Difference defined as Control minus PACESETTER at 12 months (SBP <130 mmHg); odds ratio <1 favors the PACESETTER arm

2. Secondary Outcome: Mean Systolic Blood Pressure at 12 Months
Description: Clinic systolic blood pressure (SBP, mmHg) measured at baseline, 4, 8, and 12 months after randomization. The 12-month value is reported here, comparing intervention and control arms. Lower values indicate better blood-pressure control.
Time Frame: 12 months
Population: Includes participants with at least one follow-up BP assessment (PACESETTER n=32; Control n=40). Missing values were handled using mixed-effects repeated-measures modeling under the missing-at-random assumption.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group
Number analyzed (Participants) | 32 | 40
mmHg | 132.5 (20.8) | 134.9 (18.5)
Statistical Analysis 1: Comparison: PACESETTER vs Healthy Lifestyle Intervention Group; Test type: Other — Longitudinal mixed-effects repeated-measures modeling (MMRM) was used to compare systolic BP over time, adjusting for baseline BP, site, and race; p = 0.623, Mixed Models Analysis — Two-sided α=0.05; no adjustment for multiple comparisons; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-7.3 to 12.1] — Positive values favor the control arm

3. Secondary Outcome: Mean Diastolic Blood Pressure at 12 Months
Description: Clinic diastolic blood pressure (DBP, mmHg) measured at the 12-month value is reported here, comparing intervention and control arms. Lower values indicate better blood-pressure control.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group
Number analyzed (Participants) | 32 | 40
mmHg | 85.7 (12.8) | 88 (12.1)
Statistical Analysis 1: Comparison: PACESETTER vs Healthy Lifestyle Intervention Group; Longitudinal mixed-effects repeated-measures modeling (MMRM) was used to compare diastolic BP over time, adjusting for baseline BP, site, and race; Test type: Superiority; p = 0.614, Mixed Models Analysis — Two-sided α=0.05; no adjustment for multiple comparisons; Mean Difference (Net) = -0.9, 95% CI 2-sided [-7.8 to 6.0] — Negative values favor the PACESETTER arm

ADVERSE EVENTS:
Time Frame: From randomization/enrollment until end of study follow-up at 12 months
Description: Adverse events were assessed at each study visit (baseline, 4, 8, and 12 months) using structured questionnaires and clinical evaluations. ClinicalTrials.gov definitions for adverse events were applied; no substantive differences in definitions. Analysis population includes all participants who completed at least one follow-up visit.
Arm/Group | PACESETTER | Healthy Lifestyle Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 28/60 | 21/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PACESETTER (N=60) | Healthy Lifestyle Intervention Group (N=60)
Frequent urination (nocturia) (Renal and urinary disorders) | 12 | 10
Fatigue/weakness (General disorders) | 9 | 6
Constipation/diarrhea or stool changes (Gastrointestinal disorders) | 7 | 5

LIMITATIONS AND CAVEATS:
The study did not reach the planned sample size due to COVID-19 disruptions and funding loss, resulting in high attrition and limited power. Lack of a multidisciplinary telehealth component and community-based retention strategies may have reduced engagement. Investigators and participants were unblinded, though blinded evaluators assessed outcomes. Findings may be less generalizable beyond safety-net hospitals in the Southeastern U.S.

Findings will be submitted for peer-review publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03401489/Prot_SAP_001.pdf